CLINICAL TRIAL: NCT02516644
Title: Feasibility and Effectiveness of Virtual Reality and the Use of Body Weight Support Treadmill Training in Parkinson's Disease: an Explorative Study
Brief Title: Feasibility and Effectiveness of Virtual Reality & Use of Body Weight Support Treadmill Training in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Parkinson_Xbox
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Mobility; Balance; Virtual Reality; treadmill training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual reality (Experimental): Xbox Kinect + treadmill training
  Interventions: Behavioral: Virtual Reality
- Conventional Therapy (Active Comparator): Specific conventional training for Parkinson's Disease
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: Virtual Reality — 12 sessions of 1 hour (30 min of virtual reality and 30 min of aerobic exercise with treadmill training): three times a week over four weeks
  Arms: Virtual reality
Behavioral: Conventional Therapy — 12 sessions of 1 hour of conventional physiotherapy: three times a week over four weeks
  Arms: Conventional Therapy

SUMMARY:
The primary hypothesis of the investigators is that a virtual reality system combined with physical activity provided on a body weight support treadmill training would change clinical parameters of balance and mobility in people with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson Disease diagnosis
* age under 80 years
* severity of disease rated 2 or 3 at Hoehn & Yahr scale

Exclusion Criteria:

* impaired cognitive functioning: score less than 24 on the Mini Mental State Examination
* neurologic conditions in addition to Parkinson Disease that may affect motor function and other medical conditions likely to interfere with the ability to safely complete the study protocol
* severe Levodopa dyskinesia
* pregnancy

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walking Test | up to weeks 16
  The walking endurance is measured with the Six-Minute Walking Test. Subjects are instructed to walk up and down as far as possible a 22m walkway in six minutes without encouragement, with the possibility to slow down and rest if necessary.

SECONDARY OUTCOMES:
Berg Balance Scale | weeks: 0,4, 16
  This is an assessment scale of ability to maintain balance, or statically or while performing functional movement, including 14 observable tasks common to everyday life measured on a 5 point ordinal scale.
Time Up and Go Test | weeks: 0,4, 16
  Subjects will be given verbal instruction to stand up from a chair, walk 3 meters, cross a line marked on the floor, turn around, walk back, and sit down. A study staff member will guard the subject during the test. Subjects will perform 3 trials and the time it takes to perform each trial will be recorded with a stopwatch.
10 meter walk test | weeks: 0,4, 16
  Assesses walking speed in meters per second over a short duration
Unified Parkinson's Disease Rating Scale | weeks: 0,4, 16
  It is a comprehensive assessment designed to monitor the burden and extent of Parkinson's disease across the longitudinal disease course and provide a clinical endpoint in therapy trials.
Postural sway (Center of pressure (COP) trajectories) | weeks: 0,4, 16
  Center of pressure (COP) trajectories
Metabolic measurements by Near infrared spectroscopy | weeks: 0,4, 16
  Near InfraRed Spectroscopy (NIRS) is a noninvasive, portable technique for ambulatory or remote monitoring of human motor-cortex oxygenation changes in response to motor tasks

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Principal Investigator — Ferrara Rehabilitation Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No